CLINICAL TRIAL: NCT04099732
Title: Relative Bioavailability of Rosuvastatin (Part 1) and Dabigatran (Part 2) Given Alone and Together With BI 1358894 in Healthy Male Subjects (Open, Single-dose, Fixed Sequence, Two-period Crossover Design in Each Trial Part)
Brief Title: A Study in Healthy Men to Test the Influence of BI 1358894 on the Amount of the Medicines Rosuvastatin and Dabigatran in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0009; 2019-002763-10 (EudraCT Number)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; TRPC inhibitor BI 1358894

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Reference 1 followed by Test 1 (Experimental): Reference 1 - Rosuvastatin. Test 1 - Rosuvastatin + BI 1358894
  Interventions: Drug: Rosuvastatin; Drug: BI 1358894
- Part 2: Reference 2 followed by Test 2 (Experimental): Reference 2 - Dabigatran etexilate. Test 2 - Dabigatran etexilate + BI 1358894
  Interventions: Drug: BI 1358894; Device: Dabigatran etexilate

INTERVENTIONS:
Drug: Rosuvastatin — Tablet
  Arms: Part 1: Reference 1 followed by Test 1
Drug: BI 1358894 — Tablet
Device: Dabigatran etexilate — Capsule
  Arms: Part 2: Reference 2 followed by Test 2

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of rosuvastatin (Reference 1, Part 1) and dabigatran (Reference 2, Part 2) given alone and together with BI 1358894 (Test 1, Test 2) following oral administration.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance (including positive or missing faecal occult blood test in Part 2, retest allowed)
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked prolongation of QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with women of child bearing potential (WOCBP) partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of administration of trial medication until 30 days thereafter. Sperm donation is not allowed from the time point of drug administration until 30 days thereafter.
* Known hypersensitivity to rosuvastatin or dabigatran
* Active liver disease including elevations of serum transaminases exceeding 2 times the upper limit of normal
* Moderate or severe renal impairment (creatinine clearance < 60 ml/min based on estimated Glomerular Filtration Rate (GFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Known myopathy
* Concomitant treatment with systemic cyclosporine, ketoconazole, itraconazole and dronedarone or use of fibrates
* Hypothyroidism
* Personal or family history of hereditary muscular disorders
* History of muscular toxicity with another statin or fibrate
* Asian ancestry
* Known active bleeding
* Concomitant treatment with other anticoagulants (e.g. unfractionated heparin, low molecular weight heparins, heparin derivatives, oral anticoagulants)
* Prosthetic heart valves
* Subjects who in the investigator's judgement are perceived as having an increased risk of bleeding, for example because of: current or recent gastrointestinal ulceration, presence of malignant neoplasms, recent brain or spinal injury, recent brain / spinal/ ophthalmic surgery, recent intracranial hemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms, major intraspinal or intracerebral vascular abnormalities

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open, single-dose, fixed sequence, two period crossover design to evaluate the relative bioavailability of rosuvastatin (part 1) and dabigatran (part 2) given alone and together with BI 1358894 in healthy male subjects.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that they (the subject) met all strictly implemented inclusion and None of the exclusion criteria. Subjects were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1358894 (T1): In part 1, period 1 a single oral dose of 1 film-coated tablet of 10 milligram (mg) rosuvastatin was administered with 240 milliliter (mL) of water after a high-fat, high-calorie breakfast as reference 1 (R1), followed by a washout period of at least 7 days. In part 1, period 2, a single oral dose of 1 film-coated tablet of 10 mg rosuvastatin was coadministered with a single oral dose of 2 film-coated tablets of 100 mg BI 1358894 (200 mg in total) with 240 mL of water after a high-fat, high-calorie breakfast as test 1 (T1).
- Part 2: Dabigatran (R2) / Dabigatran + BI 1358894 (T2): In part 2, period 1 a single oral dose of 1 hard capsule of 150 milligram (mg) dabigatran etexilate was administered with 240 milliliter (mL) of water after a high-fat, high-calorie breakfast as reference 2 (R2), followed by a washout period of at least 7 days. In part 2, period 2, a single oral dose of 1 hard capsule of 150 mg dabigatran etexilate was coadministered with a single oral dose of 2 film-coated tablets of 100 mg BI 1358894 (200 mg in total) with 240 mL of water after a high-fat, high-calorie breakfast as test 2 (T2).
Period: Period 1 (+ Washout Period)
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1358894 (T1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1358894 (T2)
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1358894 (T1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1358894 (T2)
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: All subjects who were entered and treated with at least 1 dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Rosuvastatin (R1) / Rosuvastatin + BI 1358894 (T1) | Part 2: Dabigatran (R2) / Dabigatran + BI 1358894 (T2) | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (7.9) | 39.7 (8.9) | 43.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 11 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 11 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part1: Area Under the Concentration-time Curve of the Analyte (Rosuvastatin) in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte (rosuvastatin) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration. Rosuvastatin + BI 1358894 (Test 1) was measured within 3 hours before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration.
Time Frame: Rosuvastatin (R1): within 3 hours before and up to 96 hours after drug administration. Rosuvastatin + BI 1358894 (1): within 3 hours before and up to 96 hours after drug administration. Detailed timeframe is provided in the description section.
Population: Pharmacokinetic (PK) parameter analysis set: All subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability
Measure: Geometric Mean (Standard Error); unit: Hours * nanogramm / milliliter
Groups:
- Rosuvastatin (Part 1, Reference 1): In part 1, period 1 a single oral dose of 1 film-coated tablet of 10 milligram (mg) rosuvastatin was administered with 240 ml of water after a high-fat, high-calorie breakfast as reference 1 (R1).
- Rosuvastatin + BI 1358894 (Part 1, Test 1): In part 1, period 2, a single oral dose of 1 film-coated tablet of 10 mg rosuvastatin was coadministered with a single oral dose of 2 film-coated tablets of 100 mg BI 1358894 (200 mg in total) with 240 mL of water after a high-fat, high-calorie breakfast as test 1 (T1).
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1358894 (Part 1, Test 1)
Number analyzed (Participants) | 14 | 14
Hours * nanogramm / milliliter | 21.19 (1.13) | 38.85 (1.13)
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1358894 (Part 1, Test 1); Relative bioavailability. The statistical model was an ANOVA model on the logarithmic scale, considering the effects 'subjects' as random and 'treatment' as fixed; Test type: Other; Ratio of geometric means (T/R) % = 183.36, 90% CI 2-sided [164.35 to 204.56] — Geometric coefficient of variation (gCV) = 16.5

2. Primary Outcome: Part 1: Maximum Measured Concentration of the Analyte (Rosuvastatin) in Plasma (Cmax)
Description: Maximum measured concentration of the analyte (rosuvastatin) in Plasma (Cmax). Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration. Rosuvastatin + BI 1358894 (Test 1) was measured within 3 hours before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration.
Time Frame: Rosuvastatin (R1): within 3 hours before and up to 96 hours after drug administration. Rosuvastatin + BI 1358894 (T1): within 3 hours before and up to 96 hours after drug administration. Detailed timeframe is provided in the description section.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Nanogramm / milliliter
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1358894 (Part 1, Test 1)
Number analyzed (Participants) | 14 | 14
Nanogramm / milliliter | 1.46 (1.14) | 2.54 (1.14)
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1358894 (Part 1, Test 1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (T/R) % = 174.01, 90% CI 2-sided [154.73 to 195.68] — Geometric coefficient of variation (gCV) = 17.7

3. Primary Outcome: Part 2: Area Under the Concentration-time Curve of the Analyte (Dabigatran) in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte (dabigatran) in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞). Dabigatran (Reference 2) was measured within 3 hours (h) before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration. Dabigatran + BI 1358894 (Test 2) was measured within 3h before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration.
Time Frame: Dabigatran (2): within 3 hours before and up to 72 hours after drug administration. Dabigatran + BI 1358894 (T2): within 3 hours before and up to 72 hours after drug administration. Detailed time frame is in description section.
Population: Pharmacokinetic (PK) parameter analysis set: All subjects included in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Deviation); unit: Hours * nanogram / milliliter
Groups:
- Dabigatran (Part 2, Reference 2): In part 2, period 1 a single oral dose of 1 hard capsule of 150 milligram (mg) dabigatran etexilate was administered with 240 ml of water after a high-fat, high-calorie breakfast as reference 2 (R2).
- Dabigatran + BI 1358894 (Part 2, Test 2): In part 2, period 2, a single oral dose of 1 hard capsule of 150 mg dabigatran etexilate was coadministered with a single oral dose of 2 film-coated tablets of 100 mg BI 1358894 (200 mg in total) with 240 mL of water after a high-fat, high-calorie breakfast as test 2 (T2).
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1358894 (Part 2, Test 2)
Number analyzed (Participants) | 12 | 12
Hours * nanogram / milliliter | 1121.67 (1.08) | 1335.96 (1.08)
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1358894 (Part 2, Test 2); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (T/R) % = 119.10, 90% CI 2-sided [109.84 to 129.15] — Geometric coefficient of variation (gCV) = 11.1

4. Primary Outcome: Part 2: Maximum Measured Concentration of the Analyte (Dabigatran) in Plasma (Cmax)
Description: Maximum measured concentration of the analyte (dabigatran) in plasma (Cmax). Dabigatran (Reference 2) was measured within 3 hours (h) before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration. Dabigatran + BI 1358894 (Test 2) was measured within 3h before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration.
Time Frame: Dabigatran (R2): within 3 hours before and up to 72 hours after drug administration. Dabigatran + BI 1358894 (T2): within 3 hours before and up to 72 hours after drug administration. Detailed time frame is in description section.
Population: as for outcome 3
Measure: Geometric Mean (Standard Error); unit: Nanogram / milliliter
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1358894 (Part 2, Test 2)
Number analyzed (Participants) | 12 | 12
Nanogram / milliliter | 112.75 (1.09) | 134.40 (1.09)
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1358894 (Part 2, Test 2); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (T/R) % = 119.20, 90% CI 2-sided [107.68 to 131.94] — Geometric coefficient of variation (gCV) = 13.9

5. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of the Analyte (Rosuvastatin) in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte (rosuvastatin) in plasma over the time interval from 0 to the last quantifiable data Point (AUC0-tz). Rosuvastatin (Reference 1) was measured within 3 hours (h) before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration. Rosuvastatin + BI 1358894 (Test1) was measured within 3 hours before drug administration and 1h, 2h, 3h, 3h 30 minutes (min) 4h, 4h 30min, 5h, 5h 30min, 6h, 7h, 8h, 10h, 12h, 24h, 34h, 48h, 72h and 96h after drug administration.
Time Frame: Rosuvastatin (R1): within 3 hours before and up to 96 hours after drug administration. Rosuvastatin + BI 1358894 (T1): within 3 hours before and up to 96 hours after drug administration. .Detailed time frame is in description section.
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: Hours * nanogram / milliliter
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1358894 (Part 1, Test 1)
Number analyzed (Participants) | 14 | 14
Hours * nanogram / milliliter | 17.56 (1.14) | 32.74 (1.14)
Statistical Analysis 1: Comparison: Rosuvastatin (Part 1, Reference 1) vs Rosuvastatin + BI 1358894 (Part 1, Test 1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (T/R) % = 186.38, 90% CI 2-sided [169.70 to 204.71] — Geometric coefficient of variation (gCV) = 14.1

6. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of the Analyte (Dabigatran) in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte (dabigatran) in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). Dabigatran (Reference 2) was measured within 3h before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration. Dabigatran + BI 1358894 (Test 2) was measured within 3h before drug administration and 1h, 1h 30min, 2h, 2h 30min, 3h, 3h 30min, 4h, 5h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration.
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) parameter analysis set: All patients included in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Hours * nanogram / milliliter
Arm/Group | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1358894 (Part 2, Test 2)
Number analyzed (Participants) | 12 | 12
Hours * nanogram / milliliter | 1086.15 (1.08) | 1304.61 (1.08)
Statistical Analysis 1: Comparison: Dabigatran (Part 2, Reference 2) vs Dabigatran + BI 1358894 (Part 2, Test 2); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (T/R) % = 120.11, 90% CI 2-sided [110.78 to 130.23] — Geometric coefficient of variation (gCV) = 11.1

ADVERSE EVENTS:
Time Frame: Adverse events occuring up to 144 hours (h) after first rosuvastatin administration in treatment period 1 of part 1 and adverse events occuring up to 168h after administration of BI 1358894 + Rosuvastatin in treatment period 2 of part 1. Adverse events occuring up to 72h after first dabigatran administration in treatment period 1 of part 2 and adverse events occuring up to 168h after administration of BI 1358894 + dabigatran in treatment period 2.
Description: Treated set: All subjects who were entered and treated with at least 1 dose of trial drug.
Groups:
- Dabigatran + BI 1355894 (Part 2, Test 2): In part 2, period 2, a single oral dose of 1 hard capsule of 150 mg dabigatran etexilate was coadministered with a single oral dose of 2 film-coated tablets of 100 mg BI 1358894 (200 mg in total) with 240 mL of water after a high-fat, high-calorie breakfast as test 2 (T2).
Arm/Group | Rosuvastatin (Part 1, Reference 1) | Rosuvastatin + BI 1358894 (Part 1, Test 1) | Dabigatran (Part 2, Reference 2) | Dabigatran + BI 1355894 (Part 2, Test 2)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/14 | 9/14 | 2/12 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin (Part 1, Reference 1) (N=14) | Rosuvastatin + BI 1358894 (Part 1, Test 1) (N=14) | Dabigatran (Part 2, Reference 2) (N=12) | Dabigatran + BI 1355894 (Part 2, Test 2) (N=12)
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 1 | 9 | 2 | 4
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04099732/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04099732/SAP_001.pdf